CLINICAL TRIAL: NCT06915311
Title: Assessment if Predictive Values of Preimplantation Genetic Testing for Aneuploidy (PGT.A). A Prospective, Blinded, Prognostic Cohort Study With the Aim of Determining if Preimplantation Genetic Testing for Aneuploidy Can be Used to Predict Clinical Outcomes.
Brief Title: Danish Prognostic Research on Embryonic Diagnostics Involving Chromosomal Testing.
Acronym: DanPREDICT
Status: Recruiting | Type: Observational
Sponsor: Christian Liebst Frisk Toft (Other)
Collaborators: Rigshospitalet, Denmark (Other); Arcedi Biotech (Industry)
Responsible Party: Sponsor-Investigator, Christian Liebst Frisk Toft, Principle Investigator, Molecular Biologist, Ph.D.,, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: N-20240008
Record Dates: First submitted 2025-04-02; First posted 2025-04-08 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Aneuploidy
Keywords: Prognostic Cohort Study; Non-selection Study; Predictive Values; Preimplantation Genetic Testing for Aneuploidy (PGT-A)
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The following samples are or might be collected as part of routine clinical care (PGT-M):
  * Embryo biopsies (5-10 trophectoderm cells removed from the blastocyst stage) [Always collected]
  * Chorionic villus sampling or amniocentesis [If patients opt for prenatal testing following PGT-M]
  The following samples are collected as part of the study:
  * Spent culture media
  * Blood sample following pregnancy for isolation of fetal cells in collaboration with ARCEDI Biotech
  * Products of conception collected following miscarriage
  * DNA sample from the newborn collected at birth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PGT-M cohort: This is the cohort on which the study will be conducted. No interventions are needed due the study design (prognostic cohort study) and the fact that embryos are already being biopsied for PGT-M.

SUMMARY:
The study aim is to evaluate whether testing embryos for chromosomal abnormalities (known as aneuploidy) can aid in embryo selection.

If so, transfer of embryos that will fail to implant, miscarry or lead to birth of affected children, can be reduces. This would reduce the risk of miscarriage and increase the chance of healthy live birth per embryo transfer, which in turn would reduce the time and economical, physical and psychological cost associated with fertility treatment.

The method of genetically testing embryos for aneuploidy is know as preimplantation genetic testing for aneuploidy (PGT-A). It entails testing a biopsy from preimplantation embryos generated from assisted reproductive technology (ART) from which DNA can be analyzed. Another potential source of embryonic DNA is the spent culture media, the media in which the embryo has grown since the egg was fertilized with the sperm. Previous research suggest that the media contains DNA shed from the embryo during development. Hence, this a potential non-invasive way of obtaining DNA for PGT-A. Both embryo biopsy and spent culture media will be assessed in the study.

The study will be conducted as a prospective, blinded, prognostic cohort study in a cohort receiving preimplantation genetic testing for monogenic disorders (PGT-M). Hence, the study does not include an intervention, as data on aneuploidy is collected but not used to guide embryo selections and embryos are biopsied as part of standard care (PGT-M). Once clinical outcomes from embryo transfers has been collected from the study, the aneuploidy data will be assessed. Blinded towards the actual clinical outcome, predictions on whether each embryo would result in live birth or not will be made based on the aneuploidy results. Following prediction, actual clinical outcomes are revealed allowing calculation of predictive values. Predictive values will be calculated for PGT-A on embryos biopsies and spent culture media.

Two predictive values will be assessed. The positive predictive value (PPV) and the negative predictive value (NPV).

The PPV states how often an embryo predicted to result in live birth upon transfer actually did so. Numerous factors affect the chance of live birth besides aneuploidy, so while the PPV will never reach 100%, it should increase compared to the PPV of standard care (without testing for aneuploidy.

The NPV states how often an embryo predicted not to result in live birth upon transfer actually also failed to do so. The NPV should be near 100 %, which would mean that all or almost all embryos that would have been deselected did not result in live birth. If the NPV is too low, it means that too many embryos capable of resulting in live birth are being discarded, disqualifying PGT-A for clinical use.

With the predictive values assessed a proper evaluation of whether PGT-A should be used clinically can be made.

A number of pre- and postnatal samples will be collected in the study to further validate PGT-A results. These include chorionic villus sampling, amniocentesis, Fetal cells isolated from maternal blood, products of conception and a DNA sample from the newborn. All of these samples can be consented to individually and as such are not required for participation in the study. Chorionic villus sampling and amniocenteses are only acquired if performed as part of routine care.

The study is expected to include 540 transfers requiring the recruitment of approximately 220 patients. Recruitment is expected to take two years combined at the two centers in Denmark participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing preimplantation genetic testing for monogenic disorders (PGT-M)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population are patients undergoing preimplantation genetic testing for monogenic disorders (PGT-M).
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | Data on live birth collected 10 months following embryo transfer.
  The primary outcome measured will be live birth rate. Positive and negative predictive values will be calculated based on the live birth rate in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Preimplantation Genetic Testing, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
It has to be investigated whether this is allowed.